CLINICAL TRIAL: NCT04855786
Title: External Drainage of Thoracic Duct Lymph to Reduce Inflammatory Cytokines in Septic Shock Patients: A Pilot Trial With Concurrent Controls to Confirm Safety and Assess Preliminary Efficacy
Brief Title: External Drainage of Thoracic Duct Lymph to Reduce Inflammatory Cytokines in Septic Shock Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Health Research Council, New Zealand (Other); University of Auckland, New Zealand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 834599
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Septic Shock
Keywords: inflammatory cytokines; Lymphatic drainage; thoracic duct; Sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thoracic Duct Drainage (Experimental): This is the main study group of patients with thoracic duct drainage
  Interventions: Procedure: Thoracic duct drainage

INTERVENTIONS:
Procedure: Thoracic duct drainage — drain placement into the thoracic duct

SUMMARY:
To demonstrate that external drainage of thoracic duct lymph during sepsis results in a reduction in circulating pro-inflammatory cytokines.

To demonstrate safety and feasibility of early thoracic duct cannulation and external lymph drainage for up to 7 days in adult surgical intensive care patients.

To explore other biochemical and physiological endpoints that can be used for the design of future randomized controlled trials and estimate effect size of external drainage.

DETAILED DESCRIPTION:
This is an interventional cohort study that will involve external drainage of thoracic duct lymph in Surgical ICU patients with septic shock. The lymph drainage will continue for up to a maximum of 7 days and will be continued in those interventional group patients discharged from ICU back to the ward before that time. The lymph (and time-matched blood) will be periodically sampled to detect changes in composition which will be correlated with changes in disease severity and outcomes, as well as patient physiology and biochemistry. This pilot study is not powered to detect changes in hospital/ICU stay, major complications or mortality. The primary endpoint of interest is the pro-inflammatory cytokine profile and concentrations in lymph and peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-80 years) patients in Surgical ICU with suspected or documented infection on antibiotics and septic shock defined as hypotension requiring vasopressor therapy to maintain MAP > 65mmHg (modified from Sepsis-35).

Participants will fulfill the inclusion criteria not only at recruitment and consent, but also be confirmed to still meet those criteria immediately prior to transfer to IR for the procedure.

The patient will not be recruited if he or she no longer meet these criteria.

Patients experiencing hemodynamic instability, defined as (1) MAPs < 65 despite ongoing up-titration of pressors and volume resuscitation or (2) active titration of vasopressors (more than 2 increases in past hour) or active volume resuscitation (more than 1-liter bolus in past hour) that precludes travel to IR during the intervention window will be excluded from the study and considered screen fails

Exclusion Criteria:

1. Open abdomen
2. Intra-abdominal sepsis preventing access to the lymphatic system
3. Prior instrumentation of the lymphatic system
4. Known occlusion of the left subclavian vein
5. Known malformation of the lymphatic system
6. Previous left axillary node dissection ± left upper limb lymphoedema
7. Class 4 heart failure
8. Any chronic medical condition for which the patient is expected to have <6-month survival
9. Decompensated liver failure with ascites
10. Portal hypertension with history of variceal bleeding
11. Severe allergy to contrast agents
12. Need for continuous anticoagulation (that cannot be stopped for procedure)
13. Uncorrectable coagulopathy or INR >1.5
14. Uncorrectable thrombocytopenia (platelet count less than 50,000)
15. Immunocompromised state (active cytotoxic chemotherapy or transplant recipient)
16. Pregnancy
17. DNR ('do not resuscitate') status
18. Subject or authorized representative not willing to provide consent (unconscious patient will need to countersign prior to analysis of samples)
19. Unable to have central venous line or arterial line in place

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in circulating pro-inflammatory cytokines | over 7 days of drainage
  serial assays of lymph and plasma to measure inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Niels D Martin, MD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No